CLINICAL TRIAL: NCT03038971
Title: A Single-Center, Double-Blinded, Placebo-Controlled, Phase 1 Evaluation of the Safety of Ragweed Mix Given in Four Monthly Doses by Intralymphatic Node Injections for Inducing Tolerance in Subjects With Ragweed Induced Allergic Conjunctivitis and Allergic Rhinitis
Brief Title: Study Evaluating Safety of Ragweed Mix Given by Intralymphatic Node Injections
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor withdrew IND from FDA
Sponsor: Woodmont Pharmaceuticals, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-290-0010
Record Dates: First submitted 2016-10-07; First posted 2017-02-01 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Allergic Conjunctivitis; Allergic Rhinitis
MeSH Terms: conditions — Conjunctivitis, Allergic; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Concentration 1: Short and Tall Ragweed Mix (Other)
  Interventions: Biological: Dose Level 1
- Concentration 2: Short and Tall Ragweed Mix (Other)
  Interventions: Biological: Dose Level 2
- Placebo: Saline with 0.4% Phenol (Other)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Dose Level 1 — Short and Tall Ragweed Mix
  Arms: Concentration 1: Short and Tall Ragweed Mix
Biological: Dose Level 2 — Short and Tall Ragweed Mix
  Arms: Concentration 2: Short and Tall Ragweed Mix
Biological: Placebo — Saline with 0.4% Phenol
  Arms: Placebo: Saline with 0.4% Phenol

SUMMARY:
A safety study conducted on subjects ≥16 years old evaluating the safety of 4 intralymphatic injections of 2 different dose levels of the investigational short and tall ragweed product. Biomarkers will be assessed at baseline and at multiple time points post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 16 and 65 years old
* Seasonal Allergic Conjunctivitis (with or without Allergic Rhinitis) to ragweed pollen
* Positive skin test reaction at screening visit to short ragweed extract
* Avoid disallowed medications
* Females of childbearing potential must have pregnancy test and must agree to use an acceptable method of birth control
* Have blood and urine analysis within normal limits
* Manifest a positive reaction to a conjunctival allergen challenge with ragweed pollen
* Have a specific IgE ≥ 0.70 kU/L to short ragweed

Exclusion Criteria:

* Have ocular or nasal conditions that could affect subject safety or trial parameters
* Have a presence of an active sinus, nasal, or ocular infections
* Have had allergy immunotherapy to ragweed pollen
* Have a compromised lung function ≤80% of predicted

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2017-04-29 (Actual); Study Completion 2017-04-29 (Actual)

PRIMARY OUTCOMES:
Adverse events (reported, elicited and observed) | 47 weeks
Local Injection Site Tolerability and Reactivity; pain will be assessed using 0-4 scale | 47 weeks
Local Injection Site Tolerability and Reactivity; tenderness will be assessed using 0-4 scale | 47 weeks
Local Injection Site Tolerability and Reactivity; redness will be assessed using 0-4 scale | 47 weeks
Local Injection Site Tolerability and Reactivity; swelling will be assessed using 0-4 scale | 47 weeks

OTHER OUTCOMES:
Conjunctival Allergen Challenge (CAC) Outcome; concentration of allergen required to elicit a positive ocular allergic reaction will be compared from baseline to 24 weeks | Baseline and up to 24 weeks
Nasal Allergen Challenge (NAC) Outcome; concentration of allergen required to elicit a positive nasal allergic reaction will be compared from baseline to 24 weeks | Baseline and up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Emily Schoemmell, Study Director — ORA, Inc.
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided